CLINICAL TRIAL: NCT03641898
Title: Intravascular Ultrasound-derived Morphometric Assessment of Fractional Flow Reserve Negative Lesions to Predict Cardiovascular Outcomes in Non-ST-segment Acute Coronary Syndrome Patients
Brief Title: Intravascular Ultrasound-derived Assessment of Hemodynamically Negative Lesions in NSTEACS Patients
Acronym: IMPACT-NSTEACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Ying Zhang, Senior Physician, Tianjin Chest Hospital
Other Study IDs: 16KG132
Record Dates: First submitted 2018-08-18; First posted 2018-08-22 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Non-ST-segment Acute Coronary Syndrome
Keywords: Fractional flow reserve; Intravascular ultrasound; Major adverse cardiovascular events; Non-ST-segment acute coronary syndrome; Percutaneous coronary intervention
MeSH Terms: interventions — Ultrasonography, Interventional

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Morphometric assessment of FNLs: After FFR-guided PCI, the morphometric characteristics of FNLs (FFR>0.8) are assessment by intravascular ultrasound.
  Interventions: Procedure: FFR-guided PCI; Diagnostic Test: Intravascular ultrasound

INTERVENTIONS:
Procedure: FFR-guided PCI — After the angiographic screening for lesions with 40%-90% diameter stenosis, FFR will be performed according to standard protocol using the s5 console and PrimeWire Prestige PLUS coronary pressure wire (Volcano Corporation, San Diego, California). FFR is calculated as the ratio of mean distal intracoronary pressure measured by the pressure wire, and the mean arterial pressure measured through the coronary guiding catheter. An FFR ≤0.8 or >90% diameter stenosis should result in a treatment decision for revascularization by PCI and lesions with FFR >0.80 are defined as FNLs and should result in deferral of PCI.
  Other Names: Functionally complete revascularization
Diagnostic Test: Intravascular ultrasound — After the successful FFR-guided PCI, IVUS will be performed in all FNLs with the ultrasound Imaging Catheter Atlantis™ SR Pro (40 MHz, mechanical-type transducer, 3.2 F, Boston Scientific Corporation, Natick, MA, USA). Quantitative analyses of grayscale IVUS include contouring external elastic membrane (EEM) and luminal borders and the measurement of EEM cross-sectional area (CSA), luminal CSA, plaque and media CSA, plaque burdenand remodeling index. Virtual assessment of plaque is performed with iMap software (QIvus 2.0; Medis Medical Imaging Systems, Leiden, The Netherlands). Plaque components are categorized as dense calcium, necrotic core, fibrofatty, and fibrous tissue and reported as absolute area and proportion of total plaque area.

SUMMARY:
This is an observational and prospective cohort study to examine whether the addition of IVUS plaque morphological evaluation to FFR haemodynamic assessment of non-culprit lesions in NSTEACS patients will better predict MACEs.

DETAILED DESCRIPTION:
IMPACT-NSTEACS is a prospective, single-centre and dynamic observational study. The study population consists of NSTEACS patients who undergo FFR in lesions with intermediate to severe angiographic stenosis. Then, FFR-guided PCI is performed, followed by morphological assessment based on IVUS in all FFR-negative lesions (FNLs). After discharge all patients receive optimal medication treatment and are followed up clinically. On the basis of follow-up angiography, MACEs are further adjudicated as occurring at FNLs or not.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Moderate to high risk NSTEACS requiring invasive strategy based on current guidelines and local clinical practice.
2. Patient agrees and is able to follow all protocol procedures.

Clinical Exclusion Criteria:

1. STEMI or SCAD.
2. Hemodynamic instability (e.g. cardiogenic shock, refractory ventricular arrhythmias, acute and severe conduction system disease and left ventricular ejection fraction ≤30%).
3. Contraindication for FFR, PCI, IVUS and OMT (e.g. severe allergy to antiplatelet drug or contrast, significant bleed within the past 6 months, bleeding diathesis and serum creatinine ≥2.5 mg/dl).
4. PCI within 6 months or any prior CABG.
5. Anticipated life expectancy <3 year.
6. Pregnancy
7. Unwilling or unable to provide informed consent

Imaging Inclusion Criteria

1. Patients must have at least > 1 de novo lesion in a native coronary segment with a visually estimated diameter stenosis of between 40 and 90 %.
2. Successful FFR-guided PCI performed in all major epicardial coronary arteries (including their branches): PCI for all lesions a) with 40%-90% diameter stenosis and FFR<0.8 and b) with ≥90% diameter stenosis.
3. The FFR-negative lesions must be available for assessment of IVUS.

Imaging Exclusion Criteria:

1. Target lesion reference diameter <2.0 mm.
2. Anatomic conditions precluding FFR and IVUS (e.g. marked calcification or tortuosity, chronic total occlusion or thrombus).
3. After successful FFR-guided PCI, no FNL is left.
4. Any remaining lesion with diameter stenosis ≥90% or FFR<0.8 after PCI.
5. Left main coronary artery lesion.
6. CABG planned by the investigators according to extent and severity of coronary artery disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For study enrollment, we screen patients with NSTEACS combination of unstable angina and non-ST-segment elevation myocardial infarction according to current guidelines. Once all clinical inclusion criteria and no clinical exclusion criteria are met, patients must sign the informed consent and undergo invasive coronary angiography (ICA). During ICA patients will be further analyzed for eligibility using angiographic inclusion and exclusion criteria. Patients will be enrolled into the study once the IVUS measurement is delivered after successful FFR-guided PCI.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The incidence and predictors of MACEs related to FNLs | 3 years
  Composite of death from cardiac causes, myocardial infarction, rehospitalization due to unstable or progressive angina and clinically-driven target lesion revascularization

SECONDARY OUTCOMES:
The incidence of MACEs related to PCI-treated lesions | 3 years
  Composite of death from cardiac causes, myocardial infarction, rehospitalization due to unstable or progressive angina and clinically-driven target lesion revascularization

OTHER OUTCOMES:
The incidence and predictors of MACEs related to FNLs | 5 years
  Composite of death from cardiac causes, myocardial infarction, rehospitalization due to unstable or progressive angina and clinically-driven target lesion revascularization
The incidence of MACEs related to PCI-treated lesions | 5 years
  Composite of death from cardiac causes, myocardial infarction, rehospitalization due to unstable or progressive angina and clinically-driven target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhang, MD, Study Chair — Tianjin Chest Hospital
Locations (1):
- Tianjin Chest Hospital, Tianjin, Tianjin Municipality, China